CLINICAL TRIAL: NCT06324045
Title: Development and Evaluation of a Multidisciplinary Team Delivered Deprescribing Intervention for Patients With Chronic Kidney Disease in Qatar: A Randomized Controlled Trial
Brief Title: Deprescribing Intervention for Patients With Chronic Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Collaborators: Qatar University (Other); Winchester District Memorial Hospital (Other)
Responsible Party: Principal Investigator, Abdullah Ibrahim Hamad, Lead Principal Investigator, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MRC-01-22-314
Record Dates: First submitted 2024-02-28; First posted 2024-03-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Diseases
Keywords: Deprescribing; Inappropriate polypharmacy; Treatment burden; Multidisciplinary; Clinical pharmacy
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Deprescriptions

STUDY DESIGN:
Intervention Model Description: CKD patients will be screened using medical records. Eligible patients will be approached during their routine visits to FBJ Kidney Center and other ambulatory kidney centers. Due to feasibility and practicality issues, selecting the patients will be consecutive case series as per their availability during the time of the recruitment (nonprobabilistic).
  After obtaining informed consent, patients will be randomized into one of the two study arms. Randomization will be stratified by dialysis dependency (dialysis vs. pre-dialysis); randomly permuted balanced block sizes of 4 for dialysis patients and 1 for pre-dialysis will be used. Neither the practitioners nor the patients will be blinded to the patients' allocated groups due to the nature of the intervention. Due to feasibility and practicalities, selecting the patients will be consecutive as per their availability during the time of the recruitment (non-probabilistic).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (No Intervention): Includes patients who will receive usual ambulatory, and at discharge care
- Intervention arm (Experimental): Includes patients who will receive a structured deprescribing intervention by the multidisciplinary team during patients' time at the center, and discharge (as applicable)
  Interventions: Other: Deprescribing

INTERVENTIONS:
Other: Deprescribing — 1. The clinical pharmacist will review the patient's medications using validated screening tools, draft a deprescribing plan of the potential problematic medications, consult with the physician (MDT-CKD nephrologist), make the needed amendments, and document in the medical records.
  2. The plan will be implemented and monitored during the patient's appointments for 1- 2 weeks at the center by the nephrologist.
  3. The medication plan will be reconciled before discharge from dialysis or a planned appointment, and patients will be given a deprescribing card containing medication information. A note will be posted on CERNER as well. The primary care physician might also be contacted by the MDT-CKD team for consultation or any inquiries regarding the patient's condition or medications.
  4. The MDT-CKD specialist nurse will conduct 3 post-appointment follow-up phone calls on day 2, day 7, and day 28 to enquire about any withdrawal symptoms or any concerns of the patient.
  Arms: Intervention arm

SUMMARY:
Chronic Kidney Disease (CKD) is recognized as a leading health problem globally. It is associated with multiple consequences such as cardiovascular diseases, infections, reduced cognitive function, and higher mortality rates. In Qatar, it is estimated that 13% of the population suffers from CKD. Management of CKD is associated with polypharmacy (the use of multiple medications), which burdens the patients and leads to adverse health and economic outcomes. As documented by previous studies, CKD setting is associated with a high medication burden, which leads to non-adherence, reduced quality of life, and other negative sequelae. These consequences can be minimized or averted by implementing a deprescribing program. Deprescribing is defined as the supervised process of intentionally stopping a medication, altering the dose or introducing a safer alternative to improve a person's clinical and quality of life outcomes. Previous deprescribing initiatives in inpatient and outpatient hospital settings were successfully implemented.

In general, there are limited deprescribing initiatives in CKD settings. There is a need to provide evidence of the impact of deprescribing programs on improving clinical and economic outcomes in this setting. In Qatar, there is no evidence of the effectiveness of implementing deprescribing programs in clinical settings. Therefore, we have built a team of researchers, clinicians, and stakeholders, and initiated a collaboration with deprescribing experts to fit into the Qatar healthcare system. This project aims to initiate a deprescribing multidisciplinary team and to evaluate the impact of providing such services on the clinical and economic outcomes among CKD patients in Qatar using a randomized controlled trial approach. The findings could have a potential positive impact on the professional practice and patient safety represented by health and economic outcomes.

DETAILED DESCRIPTION:
Medication burden and polypharmacy are evident problems among patients with CKD worldwide and in Qatar. The consequences of this problem are enormous and include high rates of adverse health and economic outcomes. Although there have been multiple initiatives to overcome polypharmacy in CKD and other chronic conditions, these initiatives still lack providing strong evidence of impact on tangible outcomes and cost-effectiveness.

In addition, most initiatives are uni-professional or fragmented. This project will initiate a multidisciplinary deprescribing program for Chronic Kidney Disease patients in Qatar. The study will also provide strong evidence of the effect of such intervention on humanistic and clinical outcomes following best practices. Undertaking deprescribing in the real world, however, is problematic; whereby, for strategic planning throughout HMC and to ensure the sustainability of the practice, including the utilization of resources and the hiring of personnel in practice sites, healthcare systems must demonstrate the return on investments made in their services. It is important, therefore, that the current study includes a cost-benefit analysis of the proposed program, to evaluate the trade-off between operational costs and the generated cost savings. The results of the study will provide an opportunity for the healthcare system in Qatar to adopt such a program among different settings that include patients prone to inappropriate polypharmacy.

Goals of the study

The goals of the proposed project are to:

1. develop and validate a deprescribing program that includes a well-trained multidisciplinary team to provide the needed care for patients with advanced stages of chronic kidney disease (CKD) who experience inappropriate polypharmacy.
2. evaluate the impact of providing a structured deprescribing program on clinical, humanistic (quality of life), and economic outcomes of advanced stages CKD patients who experience inappropriate polypharmacy.

The objectives of the study are to:

1. develop and validate an intervention framework, deprescribing guide and documents, and deprescribing training materials.
2. implement and assess the clinical and humanistic impact of the deprescribing intervention program.
3. assess the economic impact of the deprescribing intervention program on the healthcare provider institution.

The proposed project will develop and study the effect of multidisciplinary deprescribing program for patients with advanced stages of CKD and will be conducted in three consecutive phases:

* Phase I (Pre-Intervention Phase) to prepare an intervention framework and build the capacity of a multidisciplinary deprescribing team.
* Phase II (Intervention Phase) to implement and assess the clinical and humanistic impact of the deprescribing intervention program.
* Phase III (Post-Intervention Phase) to assess the economic impact of the deprescribing intervention program on the healthcare provider (i.e. HMC).

ELIGIBILITY:
Inclusion Criteria:

Patients who are:

* diagnosed with ESRD receiving hemodialysis treatment or pre-dialysis patients who are followed up at a low clearance clinic.
* receiving treatment at one of the ambulatory kidney centers in Qatar for at least two months.
* able to communicate in Arabic and/or English.

Exclusion Criteria:

* Unstable or has a psychiatric condition.
* Presents with uncontrolled behaviors or exit-seeking behaviors (i.e., seeking to leave the premises out of confusion, frustration, or anger).
* Critically ill patients, pregnant women, children, mentally ill, dementia, and unconscious patients.
* Patients with limited life expectancy (less than 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with at least one Potentially inappropriate medications (PIMs) | At baseline, 3 months, and at the end of 6 months follow-up.
  The percentage of participants with one or more PIMs. PIMs are drugs for which use should be avoided due to the high risk of adverse reactions for this population and/or insufficient evidence of their benefits when safer and equally or more effective therapeutic alternatives are available. This will be determined by outcome assessors through medical records and screening tools.
Number of Potentially inappropriate medications (PIMs) | At baseline, 3 months, and at the end of 6 months follow-up.
  The number of events and non-events in each of the study groups. PIMs are drugs for which use should be avoided due to the high risk of adverse reactions for this population and/or insufficient evidence of their benefits when safer and equally or more effective therapeutic alternatives are available. This will be determined by outcome assessors through medical records and screening tools.

SECONDARY OUTCOMES:
Pill burden | At baseline, 3 months, and at the end of 6 months follow-up.
  The frequency and total number of daily medications at baseline, and total medications that were successfully removed, dose-reduced, substituted, or restarted after intervention, categorized by targeted pharmacological drug classification.
Health-related quality of life (HRQoL) | At baseline, 3 months, and at the end of 6 months follow-up.
  This will be measured using the self-administered Kidney Disease Quality of Life (KDQOL™) questionnaire. Validated English and Arabic versions of the tool will also be used
Treatment burden | At baseline, 3 months, and at the end of 6 months follow-up.
  This will be assessed using the Treatment Burden Questionnaire (TBQ). Validated English and Arabic versions of the tool will also be used
Self-reported adherence | At baseline, 3 months, and at the end of 6 months follow-up
  The Adherence to Refills and Medications Scale (ARMS) is a validated self-administered adherence measuring tool. Validated English and Arabic versions of the tool will also be used.
Emergency department visits and hospitalizations | At baseline (indicating 6 months pre-intervention), 3 months, and at the end of 6 months follow-up.
  The total number of hospitalizations and ED visits. This will be obtained from medical records (CERNER)
Unanticipated adverse effects | At the end of 6 months follow-up
  Deprescribing is safe intervention. However, withdrawal symptoms and the need for drug re-initiation could be encountered in some cases. Each class of medications has different expected withdrawal symptoms. For example: dyspepsia after stopping PPIs. These types of events or any other unanticipated events will be documented and reported to IRB as per IRB SOP-09.
Cost avoidance | At the end of 6 months follow-up
  The cost avoided by reducing emergency department visits and hospitalization as unintended consequences of the polypharmacy use of medications. All costs will be in Qatari Riyal.
Cost savings | At the end of 6 months follow-up
  The reduced cost of therapy associated with the reduction in utilization of the targeted drugs (by deprescribing) because of the intervention program. All costs will be in Qatari Riyal.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Al-Malki, MD, Study Chair — Head of Nephrology Division, Hamad Medical Corporation; Abdullah Hamad, MD, Study Director — Division of Nephrology, Hamad Medical Corporation; Ahmed Awaisu, Ph.D., Study Director — Head of Department of Clinical Pharmacy and Practice, College of Pharmacy, Qatar University
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

REFERENCES:
- [Background] Lv JC, Zhang LX. Prevalence and Disease Burden of Chronic Kidney Disease. Adv Exp Med Biol. 2019;1165:3-15. doi: 10.1007/978-981-13-8871-2_1. PMID 31399958
- [Background] Manski-Nankervis JA, McMorrow R, Nelson C, Jesudason S, Sluggett JK. Prescribing and deprescribing in chronic kidney disease. Aust J Gen Pract. 2021 Apr;50(4):183-187. doi: 10.31128/AJGP-11-20-5752. PMID 33786539
- [Background] Johansson T, Abuzahra ME, Keller S, Mann E, Faller B, Sommerauer C, Hock J, Loffler C, Kochling A, Schuler J, Flamm M, Sonnichsen A. Impact of strategies to reduce polypharmacy on clinically relevant endpoints: a systematic review and meta-analysis. Br J Clin Pharmacol. 2016 Aug;82(2):532-48. doi: 10.1111/bcp.12959. Epub 2016 May 7. PMID 27059768
- [Background] Reeve E, Thompson W, Farrell B. Deprescribing: A narrative review of the evidence and practical recommendations for recognizing opportunities and taking action. Eur J Intern Med. 2017 Mar;38:3-11. doi: 10.1016/j.ejim.2016.12.021. Epub 2017 Jan 5. PMID 28063660
- [Background] Zidan A, Awaisu A, El-Hajj MS, Al-Abdulla SA, Figueroa DCR, Kheir N. Medication-Related Burden among Patients with Chronic Disease Conditions: Perspectives of Patients Attending Non-Communicable Disease Clinics in a Primary Healthcare Setting in Qatar. Pharmacy (Basel). 2018 Aug 13;6(3):85. doi: 10.3390/pharmacy6030085. PMID 30104554
- [Background] Al-Mansouri A, Al-Ali FS, Hamad AI, Mohamed Ibrahim MI, Kheir N, Ibrahim RA, AlBakri M, Awaisu A. Assessment of treatment burden and its impact on quality of life in dialysis-dependent and pre-dialysis chronic kidney disease patients. Res Social Adm Pharm. 2021 Nov;17(11):1937-1944. doi: 10.1016/j.sapharm.2021.02.010. Epub 2021 Feb 13. PMID 33612446
- [Background] Stewart D, Mair A, Wilson M, Kardas P, Lewek P, Alonso A, McIntosh J, MacLure K; SIMPATHY consortium. Guidance to manage inappropriate polypharmacy in older people: systematic review and future developments. Expert Opin Drug Saf. 2017 Feb;16(2):203-213. doi: 10.1080/14740338.2017.1265503. Epub 2016 Dec 4. PMID 27885844
- [Background] Kurczewska-Michalak M, Lewek P, Jankowska-Polanska B, Giardini A, Granata N, Maffoni M, Costa E, Midao L, Kardas P. Polypharmacy Management in the Older Adults: A Scoping Review of Available Interventions. Front Pharmacol. 2021 Nov 26;12:734045. doi: 10.3389/fphar.2021.734045. eCollection 2021. PMID 34899294
- [Background] Gazarin M, Devin B, Tse D, Mulligan E, Naciuk M, Duncan S, Burnett S, Hall L, Elbeddini A. Evaluating an inpatient deprescribing initiative at a rural community hospital in Ontario. Can Pharm J (Ott). 2020 Jun 9;153(4):224-231. doi: 10.1177/1715163520929734. eCollection 2020 Jul-Aug. PMID 33193924
- [Background] Ibrahim K, Cox NJ, Stevenson JM, Lim S, Fraser SDS, Roberts HC. A systematic review of the evidence for deprescribing interventions among older people living with frailty. BMC Geriatr. 2021 Apr 17;21(1):258. doi: 10.1186/s12877-021-02208-8. PMID 33865310
- [Background] Kemp A, Preen DB, Glover J, Semmens J, Roughead EE. How much do we spend on prescription medicines? Out-of-pocket costs for patients in Australia and other OECD countries. Aust Health Rev. 2011 Aug;35(3):341-9. doi: 10.1071/AH10906. PMID 21871197
- [Background] Hays RD, Kallich JD, Mapes DL, Coons SJ, Carter WB. Development of the kidney disease quality of life (KDQOL) instrument. Qual Life Res. 1994 Oct;3(5):329-38. doi: 10.1007/BF00451725. PMID 7841967
- [Background] Tran VT, Harrington M, Montori VM, Barnes C, Wicks P, Ravaud P. Adaptation and validation of the Treatment Burden Questionnaire (TBQ) in English using an internet platform. BMC Med. 2014 Jul 2;12:109. doi: 10.1186/1741-7015-12-109. PMID 24989988
- [Background] Anghel LA, Farcas AM, Oprean RN. An overview of the common methods used to measure treatment adherence. Med Pharm Rep. 2019 Apr;92(2):117-122. doi: 10.15386/mpr-1201. Epub 2019 Apr 25. PMID 31086837
- [Background] Bijlsma MJ, Janssen F, Hak E. Estimating time-varying drug adherence using electronic records: extending the proportion of days covered (PDC) method. Pharmacoepidemiol Drug Saf. 2016 Mar;25(3):325-32. doi: 10.1002/pds.3935. Epub 2015 Dec 21. PMID 26687394
- [Background] Kripalani S, Risser J, Gatti ME, Jacobson TA. Development and evaluation of the Adherence to Refills and Medications Scale (ARMS) among low-literacy patients with chronic disease. Value Health. 2009 Jan-Feb;12(1):118-23. doi: 10.1111/j.1524-4733.2008.00400.x. PMID 19911444
- [Derived] Zidan A, Hamad A, Ibrahim R, El-Kadi M, El-Malki H, Al-Esnawi M, Habib S, Abdul Hadi M, Babiker F, Al-Badriyeh D, Awaisu A. Effectiveness of a multidisciplinary team-delivered deprescribing intervention for patients with chronic kidney disease: a protocol for a randomised controlled trial. J Pharm Policy Pract. 2025 Nov 26;18(1):2588928. doi: 10.1080/20523211.2025.2588928. eCollection 2025. PMID 41358144